CLINICAL TRIAL: NCT04742075
Title: A Randomized Clinical Trial Investigating Olaparib, Durvalumab (MEDI4736) and UV1 as Maintenance Therapy in BRCAwt Patients With Recurrent Ovarian Cancer
Brief Title: Olaparib, Durvalumab and UV1 in Relapsed Ovarian Cancer
Acronym: DOVACC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: North Eastern German Society of Gynaecological Oncology (Other); Belgian Gynaecological Oncology Group (Other); Hellenic Cooperative Oncology Group (HeCOG) (Unknown); Arbeitsgemeinschaft Gynaekologische Onkologie Austria (AGO-Austria) (Unknown); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Dutch Gynaecological Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-OV56/NSGO-CTU-DOVACC
Record Dates: First submitted 2020-10-09; First posted 2021-02-05 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; durvalumab

STUDY DESIGN:
Intervention Model Description: Open-label randomized phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- (A) Olaparib (Active Comparator): Olaparib 300 mg tablets twice daily until progressive disease or unacceptable toxicity.
  Interventions: Drug: Olaparib + durvalumab + UV1
- (B) Olaparib + durvalumab (Experimental): Olaparib 300 mg tablets twice daily until progressive disease or unacceptable toxicity.
  Durvalumab 1500 mg IV every 4 weeks for 24 months or until disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib + durvalumab + UV1
- (C) Olaparib + durvalumab + UV1 (Experimental): Olaparib 300 mg tablets twice daily until disease progression or unacceptable toxicity.
  Durvalumab 1500 mg IV every 4 weeks for 24 months or until disease progression or unacceptable toxicity.
  Eight UV1 vaccinations during the first 5 month: Four UV1 vaccinations 300 μg (+ 75 μg of sargramostim) during the first 10 days with a minimum of 2 days apart. From cycle 2-5 subjects will receive one UV1 (+ sargramostim) vaccination every 4th week.
  Interventions: Drug: Olaparib + durvalumab + UV1

INTERVENTIONS:
Drug: Olaparib + durvalumab + UV1 — The subjects are randomized 1:1:2 to receive treatment until progression of disease or untorable toxicity.
  Other Names: Olaparib + durvalumab; Olaparib (active comparator)

SUMMARY:
This prospective, multicenter, open-label, randomized phase II maintenance study is evaluating the efficacy of UV1-olaparib-durvalumab combination as maintenance therapy after platinum combination therapy for BRCAwt patients with relapsed ovarian cancer.

DETAILED DESCRIPTION:
STUDY DESIGN This prospective, multicenter, open-label, randomized phase II maintenance study is evaluating the efficacy of UV1-olaparib-durvalumab combination as maintenance therapy after platinum combination therapy for BRCAwt patients with relapsed ovarian cancer.

Number of total subjects to be included in the trial:

184 patients will be enrolled in the study.

Patients are randomized into one of the three treatment arms, (A:B:C), in a 1:1:2 randomization:

* Arm A (olaparib): 46 subjects
* Arm B (olaparib plus durvalumab): 46 subjects
* Arm C (olaparib plus durvalumab plus UV1): 92 subjects

Patients are stratified according to:

* HRD status
* Previous use of PARP inhibitor (yes/no)

Primary objective:

• To compare the preliminary efficacy of maintenance treatment with olaparib (arm A) to that of olaparib plus durvalumab and UV1 (arm C)

Secondary objectives:

* To compare the preliminary efficacy of maintenance treatment with olaparib plus durvalumab (arm B) to that of olaparib plus durvalumab and UV1 (arm C)
* To compare the preliminary efficacy of maintenance treatment with olaparib plus durvalumab to that of olaparib plus durvalumab and UV1 according to stratification factors
* To evaluate Patient Reported Outcomes (PROs) in treatment arms
* To compare the preliminary efficacy of maintenance treatment according to PD-L1 status
* To evaluate safety in treatment arms

Exploratory objectives:

* To describe genetic, molecular, and immunological mechanisms in blood and tumor of maintenance treatment.
* To explore the efficacy of maintenance treatment in the molecular subgroups based on homologous recombination deficiency (HRD) status.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. The consent must be signed before the time of inclusion.
2. Histologically diagnosed with epithelial ovarian, fallopian tube or primary peritoneal cancer, excluding mucinous or low-grade serous histology.
3. Radiological or histological confirmation of relapse disease ≥ 6 months after penultimate chemotherapy.
4. Patients who are non-gBRCAmut or tBRCAwt.
5. Have completed at least two lines, but no more than 3 lines, of chemotherapy, which means that patients at first or second relapse with treatment free interval of more than 6 months on penultimate chemotherapy are eligible. See Figure 3, section 5.

   a. Patients must have completed at least 4 cycles of the latest platinum-containing chemotherapy.
6. Be either:

   1. PARPi naive.
   2. Earlier treated with PARPi and not progressed during 6 months of PARPi therapy.
7. Must not, in the opinion of the investigator, have progressed on, or after, latest platinumcontaining chemotherapy. This means that patients with CR, PR, or SD or no evidence of disease are eligible. It should be documented CR or PR on the post-treatment scan following completion of the last chemotherapy course.
8. Patient consents to HRD test (Acceptable HRD tests: Myriad myChoice® CDx, Leuven HRD test, NOGGO GISv1, and TSO 500 HRD).
9. Must be randomized in the study within 10 weeks of completion of the final dose of platinum-containing chemotherapy.
10. Age ≥18 years.
11. Body weight > 30 kg.
12. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Appendix 3)
13. Must have a life expectancy ≥ 16 weeks.
14. Must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥ 10.0 g/dL (6,2 mmol/L) with no blood transfusion in the past 28 days.
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
    * Platelet count ≥ 100 x 109/L.
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
    * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case, they must be ≤ 5x ULN.
    * Must have creatinine clearance estimated of ≥ 51 mL/min using the Cockcroft-Gault equation or based on a urine test: o Estimated creatinine clearance = [[140 - age(yr)] x weight(kg)] / [72 x serum Cr (mg/dL)] (multiply by 0.85 for women).
15. Ability to swallow oral medications (tablets) without chewing, breaking, crushing, opening, or otherwise altering the product formulation.
16. Post-menopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

Post-menopausal is defined as:

* Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments.
* Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50.
* radiation-induced oophorectomy with last menses > 1 year ago.
* chemotherapy-induced menopause with > 1 year interval since last menses.
* surgical sterilisation (bilateral oophorectomy or hysterectomy).

Exclusion Criteria:

1. Previous use of immune checkpoint inhibitors.

   a. In case the patient has participated in an immune checkpoint inhibitor blinded study, the patient may be enrolled without unblinding.
2. Other malignancy unless curatively treated with no evidence of disease for ≥ 5 years except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
3. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation ≥ 470 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
4. Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
5. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study if these were started at least 4 weeks prior to treatment.

   Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
6. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection. Examples include but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan.
7. Concomitant treatment with bevacizumab within the last 3 weeks.
8. Concomitant therapy with any other anticancer therapy or chronic use of systemic corticosteroids of more than 10mg prednisolone daily.
9. Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
10. Concomitant use of known strong CYP3A inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
11. Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation.
12. Major surgery or significant traumatic injury within 28 days of randomization.
13. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

    Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti- HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
14. Pregnancy, lactation, or intention to become pregnant during the study or/and within 1 month after the last dose of olaparib. If the patient can become pregnant, the patient must be on acceptable birth control listed in Appendix 5.
15. Participation in a clinical study within 28 days or 5 half-lives of the drug, whichever is longest.
16. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
17. Patients with a history of allergy or hypersensitivity to any of the study drugs (including human granulocyte-macrophage colony stimulating factor), yeast-derived products or any constituent of the products.
18. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy except for alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

    1. Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Sponsor.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Lead Clinician.
19. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia.
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
    3. Any chronic skin condition that does not require systemic therapy.
    4. Patients without active disease in the last 5 years may be included but only after consultation with the Sponsor.
    5. Patients with celiac disease controlled by diet alone.
20. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
21. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart). A single ECG ≥ 470 ms is sufficient.
22. History of active primary immunodeficiency.
23. Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).
24. Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP. Note:

    Patients, if enrolled, should not receive live vaccine whilst receiving IMP and up to 30 days after the last dose of IMP.
25. Has active infection with SARS-CoV-2 (antigen test).
26. Patients unable to be regularly followed for any reason (geographic, familiar, social, psychologic, housed in an institution e.g., prison because of a court agreement or administrative order according § 40 Abs. 1 S. 3 Nr. 4 AMG.).
27. Patients that are depending on the sponsor/CRO or investigational site as well as on the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 72 months
  PFS is compared between arm A versus C

SECONDARY OUTCOMES:
PFS | 72 months
  PFS is compared between arm B versus C
PFS assessed by blinded independent central review (BICR) | 72 months
  PFS is compared in each arm
Overall survival (OS) | 72 months
  OS is compared in each arm
Patient reported outcomes (PROs) - QLQ-OV28 | 72 months
  Quality of life measured by EORTC QLQ - OV28;These are the validated questionnaires to be answered by patients. Results to be reported as descriptive and on a scale of 1-10
Patient reported outcomes (PROs) - QLQ-C30 | 72 months
  Quality of life measured by EORTC QLQ - C30;These are the validated questionnaires to be answered by patients. Results to be reported as descriptive and on a scale of 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, København Ø, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Can be requested